CLINICAL TRIAL: NCT04814368
Title: A Randomized, Four-arm, Canakinumab Placebo-controlled, Participant, Investigator and Sponsor-blinded Study Investigating the Safety, Tolerability and Efficacy of Intra-articular Canakinumab Followed by Intra-articular LNA043 in Patients With Knee Osteoarthritis
Brief Title: A Safety and Efficacy Study of Anti-inflammatory (Canakinumab) and Cartilage Stimulating (LNA043) Drugs Injected Into the Knee Joint of Participants With Knee Osteoarthritis (OA)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLNA043A12203
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Results first posted 2025-07-30 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Knee Osteoarthritis
Keywords: canakinumab; LNA043; knee; osteoarthritis; OA; joint pain; cartilage; MRI; DCE-MRI; KOOS; NRS Pain; IPAQ
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Arthralgia | interventions — canakinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking only applies to the canakinumab treatment. LNA043 treatment is open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo+LNA043 (Experimental): Placebo to canakinumab on Day 1 followed by LNA043 on Days 15, 43 and 71
  Interventions: Biological: LNA043; Other: Placebo to canakinumab
- Placebo (Placebo Comparator): Placebo to canakinumab on Day 1
  Interventions: Other: Placebo to canakinumab
- canakinumab + LNA043 (Experimental): Canakinumab on Day 1 followed by LNA043 on Days 15, 43 and 71
  Interventions: Biological: canakinumab; Biological: LNA043
- canakinumab (Experimental): Canakinumab on Day 1
  Interventions: Biological: canakinumab

INTERVENTIONS:
Biological: canakinumab — Canakinumab 600 mg single intra-articular injection (into the knee) on Day 1
  Other Names: ACZ885
  Arms: canakinumab; canakinumab + LNA043
Biological: LNA043 — LNA043 40 mg intra-articular injection (into the knee) every 4 weeks, on Days 15, 43 and 71
  Arms: Placebo+LNA043; canakinumab + LNA043
Other: Placebo to canakinumab — Placebo to canakinumab single intra-articular injection (into the knee) on Day 1
  Arms: Placebo; Placebo+LNA043

SUMMARY:
The study was established to show safety and efficacy of canakinumab and LNA043 in patients with knee osteoarthritis (OA).

DETAILED DESCRIPTION:
This was a non-confirmatory, randomized, four arm, placebo-controlled, participant-, investigator and sponsor-blinded study in participants with symptomatic knee OA with synovial inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe OA pain (corresponding to NRS Pain ≥5 to ≤9) in the target knee for the majority of days in the last 3 months prior to Screening
* KOOS pain subscale <60 for the target knee during Screening
* High sensitivity C-reactive Protein (hsCRP) ≥1.8 mg/L
* Radiographic KL grade 2 to 4 knee OA and joint space width (JSW) 2.0-4.0 mm (men) or 1.5-3.5 mm (women) in the medial tibiofemoral compartment (TFC) in the target knee
* Contrast-enhanced MRI (CE-MRI) diagnosed moderate or severe knee synovitis based on an established synovititis scoring system (moderate score 9-12 or severe score ≥13)

Exclusion Criteria:

* History of, or planned; knee replacement (partial or total) in either knee; arthroscopy or lavage in either knee within 6 months prior to screening; any other previous surgical intervention in the target knee, or for the contralateral knee within 12 months prior to Screening, including mosaicplasty, microfracture, meniscectomy >50% or osteotomy
* Moderate to severe pain in the contralateral knee for the majority of days in the last 3 months prior to screening
* Malalignment >7.5° in the target knee (either varus or valgus)
* Any diagnosis of systemic inflammatory arthritis or connective tissue disease, including but not limited to rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, gout, Paget's disease, systemic lupus erythematosus) or other systemic condition that might confound assessment of OA (e.g. fibromyalgia)
* Ipsilateral hip OA or hip prosthesis recently implanted (within 1 year prior to screening) or hip replacement on either side planned within the study period

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- United States (5):
  - Horizon Clinical Research, La Mesa, California
  - Clinical Res Of W Florida, Clearwater, Florida
  - Precision Clinical Research LLC, Sunrise, Florida
  - LV Research, Las Vegas, Nevada
  - Lucas Research, Morehead City, North Carolina
- Novartis Investigative Site, Prague, Czech Republic, Czechia
- Novartis Investigative Site, Tartu, Estonia
- Hungary (2):
  - Novartis Investigative Site, Kecskemét, Bács-Kiskun county
  - Novartis Investigative Site, Budapest
- Novartis Investigative Site, Riga, Latvia
- Novartis Investigative Site, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the study in line with applicable laws and regulations.
  This study data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2679

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 11 investigative sites in 6 countries.
Pre-assignment Details: The study consisted of 4 screening visits (Screening 1-4), of which Screening 2 and 4 could be performed remotely.
Groups:
- Placebo to ACZ885+LNA043 40 mg: Placebo to ACZ885 single dose intra-articular (i.a) followed by LNA043 40 mg administrated i.a every four weeks, three times.
- Placebo to ACZ885: Placebo to ACZ885 single dose intra-articular.
- ACZ885 600 mg + LNA043 40 mg: ACZ885 600 mg single dose i.a. followed by LNA043 40 mg administrated i.a every four weeks, three times.
- ACZ885 600 mg: ACZ885 600 mg single dose intra-articular.
Period: Overall Study
Arm/Group | Placebo to ACZ885+LNA043 40 mg | Placebo to ACZ885 | ACZ885 600 mg + LNA043 40 mg | ACZ885 600 mg
Started | 3 | 9 | 3 | 8
Completed | 2 | 4 | 3 | 6
Not Completed | 1 | 5 | 0 | 2
Not completed — Study Terminated by Sponsor | 0 | 3 | 0 | 2
Not completed — Subject Decision | 1 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo to ACZ885+LNA043 40 mg | Placebo to ACZ885 | ACZ885 600 mg + LNA043 40 mg | ACZ885 600 mg | Total
Number analyzed (Participants) | 3 | 9 | 3 | 8 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (10.97) | 61.1 (5.90) | 59.3 (7.02) | 61.8 (8.55) | 61.8 (7.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 7 | 1 | 7 | 16
  Male | 2 | 2 | 2 | 1 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or other | 0 | 0 | 0 | 1 | 1
  White | 3 | 9 | 3 | 6 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Cartilage Volume in the Index Region Measured by MRI at Day 197 (Placebo to ACZ885+LNA043 Versus Placebo to ACZ885)
Description: Magnetic resonance images (MRI) were obtained from the target knee to visualize and quantify changes in volume of cartilage in the index region. The index region was defined as the union of the femoral medial anterior (FMA), central (FMC) and posterior (FMP) cartilage subregions in the knee.
Time Frame: Baseline, Day 197
Population: Participants in the pharmacodynamic (PD) analysis set from the arms "Placebo to ACZ885+LNA043 40 mg" and "Placebo to ACZ885" who had an available value for the outcome measure. The PD analysis set included all participants with available PD data and no protocol deviations with relevant impact on PD data.
Measure: Mean (Standard Deviation); unit: µL
Arm/Group | Placebo to ACZ885+LNA043 40 mg | Placebo to ACZ885
Number analyzed (Participants) | 2 | 5
µL | 108.33 (226.451) | -26.13 (65.204)

2. Primary Outcome: Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain Subscale (ACZ885 Versus Placebo to ACZ885)
Description: The KOOS questionnaire is a commonly used instrument to assess the patient's perception about their knee and associated problems. The original KOOS consists of 5 subscales. One of those is the KOOS pain consisting of 9 questions with a recall of 7days. Each question has 5 standardized answer options with a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Time Frame: Baseline, Day 85
Population: Participants in the pharmacodynamic (PD) analysis set from the arms "ACZ885 600 mg" and "Placebo to ACZ885" who had an available value for the outcome measure. The PD analysis set included all participants with available PD data and no protocol deviations with relevant impact on PD data.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | ACZ885 600 mg | Placebo to ACZ885
Number analyzed (Participants) | 8 | 7
score on scale | 22.2 (20.09) | 13.9 (13.89)

3. Secondary Outcome: Number of Participants With Anti-LNA043 Antibodies (Placebo to ACZ885+LNA043 Versus ACZ885 + LNA043)
Description: To evaluate the immunogenicity of LNA043 via validated ligand-binding assay of potential anti-LNA043 antibodies.
Time Frame: From pre-dose up to Day 365
Population: Participants in the pharmacokinetic (PK) analysis set from the arms "Placebo to ACZ885+LNA043 40 mg" and "ACZ885 600mg + LNA043 40mg" who had an available value for the outcome measure. The PK analysis set included all participants who received any study drug, and had at least one available valid (i.e. not flagged for exclusion) PK concentration measurement, and for whom there were no protocol deviations with impact on PK data.
Measure: Number; unit: Participants
Arm/Group | Placebo to ACZ885+LNA043 40 mg | ACZ885 600 mg + LNA043 40 mg
Number analyzed (Participants) | 3 | 3
Participants | 0 | 0

4. Secondary Outcome: Maximum Serum Concentration (Cmax) of ANGPTL3 (Placebo to ACZ885+LNA043 Versus ACZ885+LNA043)
Description: ANGPTL3 is a protein that is primarily involved in the lipid metabolism but has recently been shown to have chondrogenic and chondroprotective effects.
  Cmax is defined as the maximum (peak) observed concentration following a dose. ANGPTL3 serum concentrations were determined using the actual recorded sampling times and non-compartmental method with Phoenix WinNonlin (Version 8 or higher). ANGPTL3 was determined by a validated ligand binding assay; the anticipated LLOQ is 39.7 pmol/L in serum.
Time Frame: Pre-dose Day 1, Day 15, Day 43 and 60 minutes after first injection of LNA043 on Day 15
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo to ACZ885+LNA043 40 mg | ACZ885 600 mg + LNA043 40 mg
Number analyzed (Participants) | 2 | 3
ng/mL | 16.2 (2.47) | 24.1 (7.32)

5. Secondary Outcome: Synovial Fluid Concentrations of ANGPTL3 (Placebo to ACZ885+LNA043 Versus ACZ885+LNA043)
Description: ANGPTL3 is a protein that is primarily involved in the lipid metabolism but has recently been shown to have chondrogenic and chondroprotective effects.
  ANGPTL3 was measured in synovial fluid.
Time Frame: Pre-dose on Days 1, 15, 43, and 71
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo to ACZ885+LNA043 40 mg | ACZ885 600 mg + LNA043 40 mg
Number analyzed (Participants) | 1 | 1
ng/mL
  Day 1 | NA (NA) — NA = not measurable, below the lower limit of quantification of 2.74 ng/mL | NA (NA) — NA = not measurable, below the lower limit of quantification of 2.74 ng/mL
  Day 15 | NA (NA) — NA = not measurable, below the lower limit of quantification of 2.74 ng/mL | NA (NA) — NA = not measurable, below the lower limit of quantification of 2.74 ng/mL
  Day 43 | NA (NA) — NA = not measurable, below the lower limit of quantification of 2.74 ng/mL | NA (NA) — NA = not measurable, below the lower limit of quantification of 2.74 ng/mL
  Day 71 | NA (NA) — NA = not measurable, below the lower limit of quantification of 2.74 ng/mL | NA (NA) — NA = not measurable, below the lower limit of quantification of 2.74 ng/mL

6. Secondary Outcome: Maximum Serum Concentration (Cmax) of LNA043 (Placebo to ACZ885+LNA043 Versus ACZ885+LNA043)
Description: Cmax is defined as the maximum (peak) observed concentration following a dose. LNA043 serum concentrations were determined using the actual recorded sampling times and non-compartmental method with Phoenix WinNonlin (Version 8 or higher). LNA043 was determined by a validated immuno-capture and LC-MS/MS method; the anticipated LLOQ is 10 ng/mL in serum.
Time Frame: Day 15: pre-dose, 20, 60, 120 and 240 minutes, and 8 and 24 hours post LNA043 first injection on Day 15
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo to ACZ885+LNA043 40 mg | ACZ885 600 mg + LNA043 40 mg
Number analyzed (Participants) | 1 | 1
ng/mL | 120 | 149

7. Secondary Outcome: Time to Reach Maximum Serum Concentration (Tmax) of LNA043 (Placebo to ACZ885+LNA043 Versus ACZ885+LNA043)
Description: Tmax is the time to reach maximum (peak) drug concentration after single-dose administration (time). LNA043 serum concentrations were determined using the actual recorded sampling times and non-compartmental method with Phoenix WinNonlin (Version 8 or higher). LNA043 was determined by a validated immuno-capture and LC-MS/MS method; the anticipated LLOQ is 10 ng/mL in serum.
Time Frame: Day 15: pre-dose, 20, 60, 120 and 240 minutes, and 8 and 24 hours post LNA043 first injection on Day 15
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Placebo to ACZ885+LNA043 40 mg | ACZ885 600 mg + LNA043 40 mg
Number analyzed (Participants) | 1 | 1
hour | 2 | 4.02

8. Secondary Outcome: Area Under Serum Concentration-time Curve From Time Zero to the Last Measurable Concentration Sampling Time (AUClast) of LNA043 (Placebo to ACZ885+LNA043 Versus ACZ885+LNA043)
Description: AUClast is the area under the serum concentration-time curve from time zero to the time of last quantifiable concentration (tlast) of LNA043. LNA043 serum concentrations were determined using the actual recorded sampling times and non-compartmental method with Phoenix WinNonlin (Version 8 or higher). LNA043 was determined by a validated immuno-capture and LC-MS/MS method; the anticipated LLOQ is 10 ng/mL in serum.
Time Frame: Day 15: pre-dose, 20, 60, 120 and 240 minutes, and 8 and 24 hours post LNA043 first injection on Day 15
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Placebo to ACZ885+LNA043 40 mg | ACZ885 600 mg + LNA043 40 mg
Number analyzed (Participants) | 1 | 1
h*ng/mL | 800 | 1880

9. Secondary Outcome: Change in Cartilage Volume of the Index Region Measured by MRI at Day 197 and Day 365 (ACZ885+LNA043 Versus ACZ885, and ACZ885+LNA043 Versus Placebo to ACZ885+LNA043)
Description: as for outcome 1
Time Frame: Baseline, Day 197 and Day 365
Population: Participants in the pharmacodynamic (PD) analysis set from the arms "Placebo to ACZ885+LNA043 40 mg", "ACZ885 600 mg + LNA043 40 mg" and "ACZ885 600 mg" who had an available value for the outcome measure. The PD analysis set included all participants with available PD data and no protocol deviations with relevant impact on PD data.
Measure: Mean (Standard Deviation); unit: µL
Arm/Group | Placebo to ACZ885+LNA043 40 mg | ACZ885 600 mg + LNA043 40 mg | ACZ885 600 mg
Number analyzed (Participants) | 2 | 3 | 6
µL
  Day 197 | 108.33 (226.451) | 307.90 (580.213) | -82.33 (390.645)
  Day 365 | 152.78 (135.128) | 20.54 (557.708) | -129.93 (544.793)

10. Secondary Outcome: Change in Cartilage Volume of the Index Region Measured by MRI at Day 365 (Placebo to ACZ885+LNA043 Versus Placebo to ACZ885)
Description: as for outcome 1
Time Frame: Baseline, Day 365
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µL
Arm/Group | Placebo to ACZ885+LNA043 40 mg | Placebo to ACZ885
Number analyzed (Participants) | 2 | 3
µL | 152.78 (135.128) | 20.54 (557.708)

11. Secondary Outcome: Change in Cartilage Thickness of the Index Region Measured by MRI at Day 197 and Day 365 (ACZ885+LNA043 Versus ACZ885, and ACZ885+LNA043 Versus Placebo to ACZ885+LNA043)
Description: Magnetic resonance images (MRI) were obtained from the target knee to visualize and quantify changes in thickness of cartilage in the index region. The index region was defined as the union of the femoral medial anterior (FMA), central (FMC) and posterior (FMP) cartilage subregions in the knee.
Time Frame: Baseline, Day 197 and 365
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo to ACZ885+LNA043 40 mg | ACZ885 600 mg + LNA043 40 mg | ACZ885 600 mg
Number analyzed (Participants) | 2 | 3 | 7
mm
  Day 197 | 0.07 (0.083) | 0.13 (0.212) | -0.02 (0.121)
  Day 365: number analyzed (Participants) | 2 | 3 | 6
  Day 365 | -0.03 (0.046) | 0.04 (0.168) | -0.05 (0.152)

12. Secondary Outcome: Change in Cartilage Thickness of the Index Region Measured by MRI at Day 197 and Day 365 (Placebo to ACZ885+LNA043 Versus Placebo to ACZ885)
Description: as for outcome 11
Time Frame: Baseline, Day 197 and 365
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo to ACZ885+LNA043 40 mg | Placebo to ACZ885
Number analyzed (Participants) | 2 | 3
mm
  Day 197 | 0.07 (0.083) | 0.06 (0.112)
  Day 365 | -0.03 (0.046) | 0.11 (0.072)

13. Secondary Outcome: Change in Synovitis Level Measured From Ktrans by Dynamic Contrast Enhanced MRI (DCE-MRI) (ACZ885 Versus Placebo to ACZ885)
Description: Magnetic resonance images (MRI) were obtained from the target knee with dynamic contrast enhancement (DCE) to visualize and quantify changes in k-trans as a marker of the activity of synovial inflammation. During the DCE-MRI acquisition, while the contrast agent is preferentially taken up at sites with an increased perfusion due to the formation of new vessels with high porosity (such as the inflamed synovial membrane), a temporal variation of the MRI signal intensity occurs. When the contrast distributes through the intravascular and extravascular spaces, the MR signal intensity in the image volume elements (voxels) of the target tissue changes over time, generating so-called signal intensity (SI) curves. These curves can then be analyzed to derive parameters related to tissue perfusion. The parameter of primary interest was the volume transfer rate of the gadolinium-based contrast agent (GBCA) from the blood plasma in synovium, commonly referred to as Ktrans.
Time Frame: Baseline, Day 85
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: min^-1
Arm/Group | Placebo to ACZ885 | ACZ885 600 mg
Number analyzed (Participants) | 6 | 7
min^-1 | -0.0009 (0.01185) | -0.0051 (0.00702)

14. Secondary Outcome: Change in Numeric Rating Scale (NRS) Over Time (ACZ885 Versus Placebo to ACZ885)
Description: The Numerical Rating Scale (NRS) Pain is a subjective assessment in which individuals rate their pain on an eleven-point numerical scale. The scale ranges from 0 (no pain) to 10 (worst possible pain). The NRS Pain instrument had a recall period of 24 hours and the participants were asked to rate the pain intensity at its worst.
Time Frame: Baseline, Day 15, 29, 43, 57, 71, 85
Population: Participants in the pharmacodynamic (PD) analysis set from the arms "ACZ885 600 mg" and "Placebo to ACZ885" who had an available value for the outcome measure. The PD analysis set included all participants with available PD data and no protocol deviations with relevant impact on PD data. In alignment with the study protocol, data collected beyond Day 85 for NRS pain is not part of this secondary outcome measure comparing the groups ACZ885 versus Placebo to ACZ885.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo to ACZ885 | ACZ885 600 mg
Number analyzed (Participants) | 8 | 7
score on scale
  Day 15 | -1.5 (2.33) | -2.1 (2.27)
  Day 29 | -2.5 (2.73) | -3.1 (1.95)
  Day 43 | -1.8 (2.25) | -2.4 (2.15)
  Day 57: number analyzed (Participants) | 8 | 6
  Day 57 | -2.1 (2.80) | -3.5 (2.35)
  Day 71: number analyzed (Participants) | 7 | 7
  Day 71 | -2.1 (1.95) | -3.1 (2.19)
  Day 85: number analyzed (Participants) | 7 | 7
  Day 85 | -1.7 (2.29) | -2.7 (2.06)

15. Secondary Outcome: Change in Numeric Rating Scale (NRS) Over Time (ACZ885+LNA043 Versus ACZ885, and ACZ885+LNA043 Versus Placebo to ACZ885+LNA043)
Description: as for outcome 14
Time Frame: Baseline, Day 15, 29, 43, 57, 71, 85, 197 and 365
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo to ACZ885+LNA043 40 mg | ACZ885 600 mg + LNA043 40 mg | ACZ885 600 mg
Number analyzed (Participants) | 2 | 3 | 7
score on scale
  Day 15: number analyzed (Participants) | 1 | 3 | 7
  Day 15 | -3.0 | -0.7 (1.15) | -2.1 (2.27)
  Day 29: number analyzed (Participants) | 1 | 3 | 7
  Day 29 | -3.0 | -1.0 (1.00) | -3.1 (1.95)
  Day 43 | -4.5 (2.12) | -0.7 (0.58) | -2.4 (2.15)
  Day 57: number analyzed (Participants) | 1 | 3 | 6
  Day 57 | -4.0 | -2.0 (0.00) | -3.5 (2.35)
  Day 71: number analyzed (Participants) | 1 | 3 | 7
  Day 71 | -4.0 | -2.0 (1.00) | -3.1 (2.19)
  Day 85 | -5.5 (0.71) | -3.3 (0.58) | -2.7 (2.06)
  Day 197: number analyzed (Participants) | 1 | 3 | 6
  Day 197 | -6.0 | -3.3 (2.08) | -2.8 (2.64)
  Day 365: number analyzed (Participants) | 1 | 3 | 4
  Day 365 | -3.0 | -4.3 (2.31) | -3.0 (3.83)

16. Secondary Outcome: Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain Subscale Over Time (ACZ885 Versus Placebo to ACZ885)
Description: as for outcome 2
Time Frame: Baseline, Day 15, 29, 43, 57, 71, 85
Population: Participants in the pharmacodynamic (PD) analysis set from the arms "ACZ885 600 mg" and "Placebo to ACZ885" who had an available value for the outcome measure. The PD analysis set included all participants with available PD data and no protocol deviations with relevant impact on PD data. In alignment with the study protocol, data collected beyond Day 85 for KOOS pain subscale is not part of this secondary outcome measure comparing the groups ACZ885 versus Placebo to ACZ885.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo to ACZ885 | ACZ885 600 mg
Number analyzed (Participants) | 8 | 8
score on scale
  Day 15 | 12.8 (21.72) | 20.1 (20.40)
  Day 29 | 16.3 (17.60) | 24.0 (20.52)
  Day 43 | 11.8 (12.31) | 21.9 (21.28)
  Day 57 | 13.9 (18.96) | 28.1 (19.38)
  Day 71: number analyzed (Participants) | 7 | 8
  Day 71 | 14.3 (15.75) | 26.4 (20.03)
  Day 85: number analyzed (Participants) | 7 | 8
  Day 85 | 25.0 (3.93) | 22.2 (20.09)

17. Secondary Outcome: Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain Subscale Over Time (ACZ885+LNA043 Versus ACZ885, and ACZ885+LNA043 Versus Placebo to ACZ885+LNA043)
Description: as for outcome 2
Time Frame: Baseline, Day 15, 29, 43, 57, 71, 85, 197 and 365
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo to ACZ885+LNA043 40 mg | ACZ885 600 mg + LNA043 40 mg | ACZ885 600 mg
Number analyzed (Participants) | 2 | 3 | 8
score on scale
  Day 15 | 25.0 (27.50) | 3.7 (18.91) | 20.1 (20.40)
  Day 29 | 36.1 (19.64) | 15.7 (9.76) | 24.0 (20.52)
  Day 43 | 25.0 (15.71) | 15.7 (16.74) | 21.9 (21.28)
  Day 57 | 25.0 (7.86) | 17.6 (5.78) | 28.1 (19.38)
  Day 71 | 29.2 (5.89) | 16.7 (2.78) | 26.4 (20.03)
  Day 85 | 25.0 (3.93) | 22.2 (14.70) | 22.2 (20.09)
  Day 197 | 37.5 (9.82) | 38.0 (12.83) | 25.0 (21.87)
  Day 365: number analyzed (Participants) | 2 | 3 | 6
  Day 365 | 31.9 (17.68) | 45.4 (10.52) | 31.5 (26.33)

18. Secondary Outcome: Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) Function in Daily Living (ADL) Subscale Over Time (ACZ885 Versus Placebo to ACZ885)
Description: The KOOS questionnaire is a commonly used instrument to assess the patient's perception about their knee and associated problems. The original KOOS consists of 5 subscales. One of those is the KOOS Function in Daily Living (ADL) subscale consisting of 17 questions with a recall of 7days. Each question has 5 standardized answer options with a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Time Frame: Baseline, Day 15, 29, 43, 57, 71, 85
Population: Participants in the pharmacodynamic (PD) analysis set from the arms "ACZ885 600 mg" and "Placebo to ACZ885" who had an available value for the outcome measure. The PD analysis set included all participants with available PD data and no protocol deviations with relevant impact on PD data. In alignment with the study protocol, data collected beyond Day 85 for KOOS function in daily living subscale is not part of this secondary outcome measure comparing the groups ACZ885 versus Placebo to ACZ885.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo to ACZ885 | ACZ885 600 mg
Number analyzed (Participants) | 8 | 8
score on scale
  Day 15 | 11.9 (23.87) | 18.4 (18.35)
  Day 29 | 14.3 (24.74) | 25.7 (20.72)
  Day 43 | 9.7 (17.04) | 26.1 (19.79)
  Day 57 | 16.7 (28.06) | 31.8 (21.99)
  Day 71: number analyzed (Participants) | 7 | 8
  Day 71 | 16.8 (22.30) | 28.7 (19.40)
  Day 85: number analyzed (Participants) | 7 | 8
  Day 85 | 14.7 (23.05) | 23.7 (19.26)

19. Secondary Outcome: Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) Function in Daily Living (ADL) Subscale Over Time (ACZ885+LNA043 Versus ACZ885, and ACZ885+LNA043 Versus Placebo to ACZ885+LNA043)
Description: as for outcome 18
Time Frame: Baseline, Day 15, 29, 43, 57, 71, 85, 197 and 365
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo to ACZ885+LNA043 40 mg | ACZ885 600 mg + LNA043 40 mg | ACZ885 600 mg
Number analyzed (Participants) | 2 | 3 | 8
score on scale
  Day 15 | 37.5 (34.32) | 2.9 (8.82) | 18.4 (18.35)
  Day 29 | 42.6 (20.80) | 17.2 (4.49) | 25.7 (20.72)
  Day 43 | 41.9 (28.08) | 16.2 (11.76) | 26.1 (19.79)
  Day 57 | 40.4 (19.76) | 19.1 (8.95) | 31.8 (21.99)
  Day 71 | 43.4 (23.92) | 20.6 (10.29) | 28.7 (19.40)
  Day 85 | 41.9 (19.76) | 28.4 (15.09) | 23.7 (19.26)
  Day 197 | 50.7 (19.76) | 36.8 (1.47) | 27.4 (23.92)
  Day 365: number analyzed (Participants) | 2 | 3 | 6
  Day 365 | 44.9 (26.00) | 42.2 (13.34) | 33.6 (23.79)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus follow up period, up to a maximum duration of approximately 52 weeks.
Groups:
- Total: Total
Arm/Group | Placebo to ACZ885+LNA043 40 mg | Placebo to ACZ885 | ACZ885 600 mg + LNA043 40 mg | ACZ885 600 mg | Total
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/9 | 0/3 | 0/8 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/9 | 0/3 | 0/8 | 0/23
Other Adverse Events (participants affected / at risk) | 1/3 | 2/9 | 1/3 | 4/8 | 8/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo to ACZ885+LNA043 40 mg (N=3) | Placebo to ACZ885 (N=9) | ACZ885 600 mg + LNA043 40 mg (N=3) | ACZ885 600 mg (N=8) | Total (N=23)
Bundle branch block right (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Body tinea (Infections and infestations) | 0 | 1 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1

LIMITATIONS AND CAVEATS:
The small sample size overall and the difference in group sizes do not allow a valid interpretation of the data regarding efficacy, pharmacokinetics and immunogenicity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT04814368/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT04814368/SAP_001.pdf